CLINICAL TRIAL: NCT03821142
Title: Prospective, Multicenter, 60 Months, Single Arm Cohort Study to Evaluate the Efficacy and Safety of the Ultra-Light-Weight Mesh CAlistar S in Transvaginal Pelvic Organ Prolapse Repair
Brief Title: Prospective Long-term Evaluation of the Efficacy and Safety of Calistar S for Transvaginal Pelvic Organ Prolapse Repair
Acronym: CASPO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Promedon (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CaS_Pro
Record Dates: First submitted 2019-01-10; First posted 2019-01-29 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Pelvic Organ Prolapse
Keywords: surgical mesh; surgery; Therapy; pelvic floor disorders; cystocele
MeSH Terms: conditions — Pelvic Organ Prolapse; Pelvic Floor Disorders; Cystocele

STUDY DESIGN:
Intervention Model Description: Calistar S Single Incision POP System
Masking Description: Blinded POP-Q Examination: The POP-Q examination will be performed by a physician different to the corresponding surgeon
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Calistar S (Experimental): Single arm cohort trial
  Interventions: Device: Transvaginal mesh for anterior pelvic organ prolapse repair

INTERVENTIONS:
Device: Transvaginal mesh for anterior pelvic organ prolapse repair — synthetic mesh for anterior pelvic organ prolapse with or without apical vaginal wall involvement via the vaginal route in a highly selected patient population

SUMMARY:
Prospective long-term evaluation of the performance and safety of Calistar S for transvaginal pelvic organ prolapse repair in women with anterior POP with or without apical vaginal involvement

DETAILED DESCRIPTION:
Calistar S Single Incision Pelvic Organ Prolapse (POP) Repair System is intended for transvaginal reestablishment and reinforcement of the physiologic anatomy of the female pelvic floor in non-fertile women with anterior pelvic organ prolapse with or without apical vaginal wall involvement in both, recurrent pelvic organ prolapse and primary pelvic organ prolapse when other surgical procedures are expected to fail (i.e. complex primary prolapse).

The treatment kit consists of the lightweight mesh, two single-use introducers and 3 tissue anchoring system (TAS) anchors for fixation to the sacrospinous ligament. The product is approved in accordance with the CE Directive 93/42/EEC.

The utilization of synthetic implants in POP repair became increasingly popular in the last decade. The cumulative success rate of synthetic implants in anterior compartment repair is as high as up to 93%.However, meshes have been recently scrutinized due to high adverse event reporting after unreflected utilization of meshes which raised concerns of patients safety; furthermore taking into account the complexity of adverse event mesh management. This led to a vanishing of various meshes in transvaginal POP repair. Nevertheless, the further development of light weight meshes, the experience of the surgeon and the assessment and patients selection are well known factors reducing the rate of adverse events significantly.

Therefore, in the current trial the efficacy and safety of calistar S in a highly selected patient population will be evaluated.

ELIGIBILITY:
Inclusion criteria Non-fertile women > 18 years1 2. Symtomatic anterior prolapse with or without apical vaginal wall involvement according POP-Q score ≥ 2. (Corresponding to Aa, Ba ≥ -1 and where applicable C ≥ -1/2 TVL ).

3. Subjects with recurrent prolapse or complex primary prolapse are eligible for the study.

4. Scheduled mesh-augmented anterior POP repair with Calistar S 5. Signed inform consent

Exclusion criteria

1. Fertile women
2. Patients with active or latent infection of the vagina, cervix or uterus
3. Patients with previous or current vaginal, cervical or uterine cancer
4. Previous, current or planned pelvic radiation therapy
5. Known allergy to polypropylene

7. Subject is unable or unwilling to complete questionnaires (either self-administered, assisted or interviewed) and/or to follow scheduled visits and/or to sign informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2021-03-10 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Number of Patients with Cure of pelvic organ prolapse | 24 months
  Number of patients accomplishing the composite endpoint after 24 months including anatomic, subjective and retreatment components

SECONDARY OUTCOMES:
Change of prolapse specific quality of life according the validated Questionnaire Prolapse quality of life questionnaire in comparison between baseline and follow-up | Baseline, 6 weeks and 6, 12, 24, 36, 48, 60 months
  Differences between Baseline and Follow-Up result of the questionnaire of each patient regarding Quality of life and the correlating domains will be evaluated. P-QoL, Score: 0-100, the higher the score, the higher the impact of prolapse symptoms and the lower quality of life.
Change of sexual life according the Pelvic Organ Prolapse/Incontinence Sexual Questionnaire in comparison between Baseline and follow-up | Baseline, 6 weeks and 6, 12, 24, 36, 48, 60 months
  Differences between Baseline and Follow-Up result of each patient regarding Sexual life and the correlating domains will be evaluated. PISQ-IR, Score: 0-100, the higher the score, the higher the impact of prolapse symptoms and the higher the impact on sexual life.
Change of pain according Visual Analog Scale of Pain in comparison between baseline, postoperative and follow-up | Baseline, 24-48h postoperatively, 6 weeks and 6, 12, 24, 36, 48, 60 months
  Differences of pain-evaluation between Baseline and Follow-Up of each patient will be evaluated. Wong Baker Pain Scale, Score: 0 - 10, The higher the score, the higher the pain.
Patients subjective evaluation of satisfaction with surgery according the Patient Global Impression of Improvement | 6 weeks and 6, 12, 24, 36, 48, 60 months
  Evaluation of the improvement of POP after the operation assed by the Patient Global Impression of Improvement of each patient. PGI-I, Score: 7 Likert scale from: very much better to very much worse,
Patient subjective evaluation of POP severity according the Global Impression of Severity | Baseline
  Evaluation of severity categorization by assing the Patient Global Impression of Severity of each patient at Baseline. Score. 4 Likert scale, from no impact to very much impact. A
Change of quality of life according the EQ-5L-5D in comparison between baseline and follow-up | Baseline, 6 weeks and 6, 12, 24, 36, 48, 60 months
  Evaluation of Quality of life assessed by the EQ-5L-5D and evaluation of differences between Baseline and Follow-Up of each patient regarding health related Quality of life. Two scores: a) 5 Likert scale from no problems to extreme problems. b) self administered quality of life in scale 0 - 100, the higher the score the better the quality of life.
Anatomical success according the number of patients with anterior vaginal wall at or above the hymen and no decent of apical vaginal wall at or greater than half of the total vanilla lengths | 6 weeks and 6, 12, 24, 36, 48, 60 months
  Anatomical success defined by the number of patients with the anterior vaginal wall at or above the hymen (Aa and Ba ≤ 0 ) and separately no decent of apical vaginal wall at or greater than half of the total vaginal lengths (C < -½ TVL).
Number of patients with necessity of repeated surgery due to recurrent anterior or apical Number of patients with Repeat surgery due to symptomatic recurrence of anterior or apical POP | 6 weeks and 6, 12, 24, 36, 48, 60 months
  Number of patients with necessity of repeated surgery due to recurrent anterior or apical POP.
Safety of Calistar S according the number of adverse events | intraoperative, postoperative, 6 weeks, and 6, 12, 24, 36, 48, 60 months and unscheduled visits
  Safety of Calistar S according the assessment of total amount of adverse events
Exposure and anatomical-failure free survival | 12, 24, 36, 48, 60 months
  Estimation of exposure- and anatomical-failure free survival according Kaplan meier
Number of patients with further surgery for stress urinary incontinence | 6 weeks and 6, 12, 24, 36, 48, 60 months
  To assess the number of patients with further surgery for stress urinary incontinence.
Change of urinary incontinence according the ICIQ-UI-Sf in comparison between baseline and follow-up | Baseline 6 weeks and 6, 12, 24, 36, 48, 60 months
  The international Consultation of Incontinence Questionnaire - Urinary Incontinence - Short Form (ICIQ-UI-SF) is a validated questionnaire to asses urinary incontinence. Score 0-21, overall score with greater values indicating increased symptom severity
Change of overactive bladder symptoms according the ICIQ-OAB in comparison between baseline and follow-up | Baseline 6 weeks and 6, 12, 24, 36, 48, 60 months
  The International Consultation of Incontinence Questionnaire - Overacitve bladder (ICIQ-OAB) is a validated questionnaire.. 0-16 overall score with greater values indicating increased symptom severity
Cure in short-, mid-, and longterm follow-up | 6 weeks and 6, 12, 36, 48, 60 months
  Number of patients accomplishing the composite outcome at remaining follow-up times

CONTACTS AND LOCATIONS:
Overall Officials: Gert Naumann, PD Dr.habil., Principal Investigator — Helios Hospital Erfurt; Ralf Tunn, Prof.Dr., Principal Investigator — St. Hedwig Hospital; Dirk Watermann, Prof.Dr., Principal Investigator — Evangelic Diakonie Hospital; Birgit Henne, Dr.med., Principal Investigator — St. Elisabeth-Hospital Leipzig; Christl Reisenauer, Prof.Dr.med., Principal Investigator — University Hospital Tübingen; Christian Fünfgeld, Dr.med., Principal Investigator — Hospital Tettnang
Locations (6):
- Germany (6):
  - Helios Hospital Erfurt, Department of gynaecology, Erfurt, Thuringia
  - St. Hedwig Hospital, Berlin
  - Evangelic Diakonie Hospital, Freiburg im Breisgau
  - St. Elisabeth-Hospital Leipzig, Leipzig
  - Hospital Tettnang, Tettnang
  - University Hospital Tübingen, Tübingen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Olsen AL, Smith VJ, Bergstrom JO, Colling JC, Clark AL. Epidemiology of surgically managed pelvic organ prolapse and urinary incontinence. Obstet Gynecol. 1997 Apr;89(4):501-6. doi: 10.1016/S0029-7844(97)00058-6. PMID 9083302
- [Background] Wu JM, Matthews CA, Conover MM, Pate V, Jonsson Funk M. Lifetime risk of stress urinary incontinence or pelvic organ prolapse surgery. Obstet Gynecol. 2014 Jun;123(6):1201-1206. doi: 10.1097/AOG.0000000000000286. PMID 24807341
- [Background] Wu JM, Vaughan CP, Goode PS, Redden DT, Burgio KL, Richter HE, Markland AD. Prevalence and trends of symptomatic pelvic floor disorders in U.S. women. Obstet Gynecol. 2014 Jan;123(1):141-148. doi: 10.1097/AOG.0000000000000057. PMID 24463674
- [Background] Hendrix SL, Clark A, Nygaard I, Aragaki A, Barnabei V, McTiernan A. Pelvic organ prolapse in the Women's Health Initiative: gravity and gravidity. Am J Obstet Gynecol. 2002 Jun;186(6):1160-6. doi: 10.1067/mob.2002.123819. PMID 12066091
- [Background] Mant J, Painter R, Vessey M. Epidemiology of genital prolapse: observations from the Oxford Family Planning Association Study. Br J Obstet Gynaecol. 1997 May;104(5):579-85. doi: 10.1111/j.1471-0528.1997.tb11536.x. PMID 9166201
- [Background] Risk factors for genital prolapse in non-hysterectomized women around menopause. Results from a large cross-sectional study in menopausal clinics in Italy. Progetto Menopausa Italia Study Group. Eur J Obstet Gynecol Reprod Biol. 2000 Dec;93(2):135-40. PMID 11074133
- [Background] Barber MD, Kuchibhatla MN, Pieper CF, Bump RC. Psychometric evaluation of 2 comprehensive condition-specific quality of life instruments for women with pelvic floor disorders. Am J Obstet Gynecol. 2001 Dec;185(6):1388-95. doi: 10.1067/mob.2001.118659. PMID 11744914
- [Background] Barber MD, Walters MD, Bump RC. Short forms of two condition-specific quality-of-life questionnaires for women with pelvic floor disorders (PFDI-20 and PFIQ-7). Am J Obstet Gynecol. 2005 Jul;193(1):103-13. doi: 10.1016/j.ajog.2004.12.025. PMID 16021067
- [Background] Lenz F, Stammer H, Brocker K, Rak M, Scherg H, Sohn C. Validation of a German version of the P-QOL Questionnaire. Int Urogynecol J Pelvic Floor Dysfunct. 2009 Jun;20(6):641-9. doi: 10.1007/s00192-009-0809-x. Epub 2009 Feb 13. PMID 19214361
- [Background] Digesu GA, Khullar V, Cardozo L, Robinson D, Salvatore S. P-QOL: a validated questionnaire to assess the symptoms and quality of life of women with urogenital prolapse. Int Urogynecol J Pelvic Floor Dysfunct. 2005 May-Jun;16(3):176-81; discussion 181. doi: 10.1007/s00192-004-1225-x. Epub 2004 Oct 21. PMID 15875234
- [Background] Rogers RG, Coates KW, Kammerer-Doak D, Khalsa S, Qualls C. A short form of the Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ-12). Int Urogynecol J Pelvic Floor Dysfunct. 2003 Aug;14(3):164-8; discussion 168. doi: 10.1007/s00192-003-1063-2. Epub 2003 Jul 25. PMID 12955337
- [Background] Wong DL, Baker CM. Smiling faces as anchor for pain intensity scales. Pain. 2001 Jan;89(2-3):295-300. doi: 10.1016/s0304-3959(00)00375-4. No abstract available. PMID 11291631
- [Background] Bump RC, Mattiasson A, Bo K, Brubaker LP, DeLancey JO, Klarskov P, Shull BL, Smith AR. The standardization of terminology of female pelvic organ prolapse and pelvic floor dysfunction. Am J Obstet Gynecol. 1996 Jul;175(1):10-7. doi: 10.1016/s0002-9378(96)70243-0. PMID 8694033
- [Background] Vittinghoff E, McCulloch CE. Relaxing the rule of ten events per variable in logistic and Cox regression. Am J Epidemiol. 2007 Mar 15;165(6):710-8. doi: 10.1093/aje/kwk052. Epub 2006 Dec 20. PMID 17182981
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Practice Bulletin No. 176: Pelvic Organ Prolapse. Obstet Gynecol. 2017 Apr;129(4):e56-e72. doi: 10.1097/AOG.0000000000002016. PMID 28333818